CLINICAL TRIAL: NCT01863719
Title: A Phase 1, Open-Label Study of the Safety, Tolerability and Pharmacokinetics of Aerosolized Colistimethate Sodium After Multiple Doses Administered Separately or in Combination With Intravenous Colistimethate Sodium in Healthy Adults
Brief Title: Aerosolized and Intravenous Colistin in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Completion of cohort 3, safety concerns
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0082; HHSN272201500007I
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02-25

CONDITIONS: Pathogen Resistance; Pneumococcal Infection; Pneumonia
Keywords: Colistin; Multi Drug Resistant; Nosocomial Pneumonia; Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia; Healthcare-Associated Pneumonia | interventions — colistinmethanesulfonic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): 9 Subjects
  Interventions: Drug: Colistimethate sodium
- Cohort 2 (Experimental): 9 Subjects
  Interventions: Drug: Colistimethate sodium
- Cohort 3 (Experimental): 9 Subjects
  Interventions: Drug: Colistimethate sodium
- Cohort 4 (Experimental): 12 Subjects
  Interventions: Drug: Colistimethate sodium

INTERVENTIONS:
Drug: Colistimethate sodium — Aerosol: In Dosing period 2 subjects receive 75mg colistin base activity via aerosol every 6 hours x 4 doses, followed by a washout period of at least 3 days. In Dosing period 3 subjects receive 75mg colistin base activity via aerosol every 6 hours x 4 doses in combination with 3.3mg/kg colistin base activity IV every 8 hours x 3 doses.
Drug: Colistimethate sodium — Intravenous: In Dosing period 1 subjects receive 3.3mg/kg colistin base activity every 8 hours x 3 doses (total exposure 10mg/kg) intravenously (IV) followed by a washout period of at least 3 days. In Dosing period 3 subjects receive 3.3mg/kg colistin base activity IV every 8 hours x 3 doses in combination with 75mg colistin base activity via aerosol every 6 hours x 4 doses.

SUMMARY:
Colistin is amphipathic, cannot be absorbed from the gastrointestinal tract and is administered intramuscularly, intravenously (IV) or via inhalation. In the case of pneumonia, aerosolized route of administration is favorable as it presumably delivers a high concentration of drug directly to the infection site. Colistimethate sodium is an FDA approved drug, however, its aerosolized use represents a new method of administration not currently FDA-approved in the United States. In this proposal, the inactive prodrug colistimethate sodium has been selected to use for aerosolization as it is better tolerated than colistin sulphate. It is a randomized, open-labeled Phase 1 trial of aerosolized and/or IV formulations of colistin as multiple doses over seven days. The primary objective of this trial is to evaluate the safety and tolerability of multiple doses of aerosolized and intravenous colistimethate sodium separately or in combination in healthy adult subjects.

DETAILED DESCRIPTION:
"Colistin" (the first breakdown product colistimethate sodium, also known as polymyxin E) is comprised of approximately 30 different polymyxins, with colistin A (polymyxin E1) and colistin B (polymyxin B) accounting for upwards of 85% of the mass. It is amphipathic, cannot be absorbed from the gastrointestinal tract and is administered intramuscularly, intravenously (IV) or via inhalation. While approved for aerosolized use in the United Kingdom, and used in Europe for decades as such, aerosolized colistin is not FDA-approved in the United States. The intravenous formulation is approved for use in the U.S., but due to the age of the drug, it did not undergo rigorous studies of safety prior to FDA-approval. Thus, detailed pharmacokinetic data are limited and dosing is not standardized, although the maximum IV dose should not exceed 5mg/kg/day, divided into two to four equal doses. In the United Kingdom, the recommended dosing of nebulized colistin for adults is one million units (1MIU) twice daily. Despite the paucity of dosing and safety guidelines, aerosolized colistin is being prescribed regularly out of necessity given the emergence of multi-drug resistant organisms (MDROs). MDROs are strongly associated with nosocomial pneumonia and several strains are only susceptible to this older drug, thus there is an urgent need for clarification on the safe use of colistin, including in aerosolized form as this delivers a high concentration of drug directly to the infection site. This is a randomized, open-labeled Phase 1 trial of aerosolized and/or IV formulations of colistin as multiple doses over seven days. 39 healthy male and female subjects, 18-45 years of age will be admitted for an inpatient study with outpatient follow-up. The primary objective of this trial is to evaluate the safety and tolerability of multiple doses of aerosolized and intravenous colistimethate sodium separately or in combination in healthy adult subjects. The secondary objective of this trial is to determine the pharmacokinetics of multiple daily doses of aerosolized and intravenous colistimethate sodium separately or in combination in healthy adult subjects. Subjects will participate for up to 25 days plus a screening and a follow-up appointment. The duration of this study shall be for two years, including screening, study conduct (including scheduled SMC reviews), study follow-up and preparation of all reports.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained and signed 2. Aged between 18 and 45 years, inclusive 3. Body Mass Index (BMI, weight in kg divided by the square of height in meters) between 18 and 35.0 kg/m^2, inclusive 4. Able to comply with protocol requirements for the entire duration of the study 5. Healthy on the basis of a screening medical evaluation (including physical examination, vital signs, blood biochemistry and hematology, urinalysis, and history).

Exclusion Criteria:

1. Heterosexually active females of child-bearing potential, defined as being physiologically capable of becoming pregnant, unless they agree to use two of the following acceptable methods of contraception throughout their participation in the study and for at least 12 weeks after the final dose: (a) established use of oral, injected or implanted hormonal contraception, (b) intrauterine Device (IUD or Coil) (c) a female barrier method (diaphragm or cervical/vault cap) and/or (d) condom plus spermicidal cream/gel 2. Heterosexually active males unless they agree to use two concomitant acceptable methods of contraception throughout their participation in the study and for at least 12 weeks after receiving their final dose of study medication (examples include: vasectomy combined with latex condom with spermicide, latex condom with spermicide combined with a female partner who practices an acceptable method of contraception as indicated above) 3. History or current abuse of alcohol, barbiturates, amphetamines, tetrahydrocanninol, phencyclidine, cocaine, heroin, or other narcotics, as evidenced by a reported history or positive screen for these agents 4. Any clinically significant (as deemed by the Principal Investigator) history of asthma; cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (including eating disorders), endocrine, metabolic, immunologic, dermatologic, neurologic (including a history of seizures, ataxia, or Myastenia Gravis), psychological, or psychiatric disease; and/or a past or family history of porphyria 5. Use of tobacco/nicotine within 3 months prior to Screening and for the entire duration of the study); 6. Treatment with another investigational drug 60 days prior to and/or during the study 7. Co-enrollment in another study involving the intake of medication 8. Immunocompromised status, including a positive HIV-1 (Human Immunodeficiency Virus) or HIV-2 test by ELISA at screening 9. Previously demonstrated clinically significant allergy or hypersensitivity to colistimethate sodium or its excipients 10. Donation of blood or significant blood loss within 56 days of study Enrollment or during study duration, or plasma donation within 28 days preceding study Enrollment 11. Hepatitis B, or C infection (confirmed by hepatitis B surface antigen, or hepatitis C virus antibody, respectively) at screening 12. Laboratory abnormalities at Screening as outlined below: a. Serum creatinine (>/=1.1 x ULN), b. Hemoglobin (<11.0 or >17.5g/dL), c. Platelet count (<125,000 or >450,000/mm^3), d. Absolute neutrophil count (<1300mm^3), e. Serum blood urea nitrogen (>/=1.2 x ULN) f. Aspartate aminotransferase (AST, >/=1.2 x ULN), g. Alanine aminotransferase (ALT, >/=1.2 x ULN), h. Proteinuria (spot urine) greater than trace and/or hematuria greater than trace; Note: Subjects may undergo a repeat screening test of out-of-range analyte(s) at the discretion of the investigator to confirm a plausible alternative explanation that will be indicated in the source documentation. A repeat laboratory test may be used to satisfy eligibility requirements. 13. Intake of any of the following medications within 30 days prior to Screening and during the study: acyclovir, adefovir, aminoglycosides, amphotericin, cisplatin, cyclosporine, fluoroquinolones, foscarnet, ganciclovir, pamidronate, sirolimus, tacrolimus, and vancomycin, and/or any neuromuscular blockers;- Intake of NSAIDs (ibuprofen, naproxen, etodolac) within 48 hours of dosing and any inhaled medication within 5 days of dosing. Additionally, subjects may be excluded due to intake of medications not listed here at the discretion of the PIs (Principal Investigators) 14. Intake of NSAIDs (ibuprofen, naproxen, etodolac) within 48 hours of dosing and any inhaled medication within 5 days of dosing. Additionally, subjects may be excluded due to intake of medications not listed here at the discretion of the PIs; 15. FEV1 (Forced Expiratory Volume) <80 percent predicted 16. Prior evidence (symptoms within the past year) of vestibular problems or neuropathy 17. Abnormal QT interval at screening ECG (Electrocardiogram) (Bazett correction >450 milliseconds) or significant abnormities according to the cardiologist's final reading 18. A grade 3 or 4 clinical or confirmed laboratory toxicity (as outlined in Appendix C) which does not return to grade 2 or lower; 19. Any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk or injury, or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
The occurrence of solicited and unsolicited adverse events, including symptoms, physical findings, laboratory testing (hematology, chemistries, urinalysis), and ECG changes | Enrollment through to 2 weeks after end of dosing period 3

SECONDARY OUTCOMES:
Pharmacokinetic effect of colistimethate sodium: measure of bronchoalveolar lavage (BAL) colistimethate sodium, colistin A, and colistin B levels. | BAL: 3hrs after completion of each dose, (in 3 of 9 subjects per cohort)
Pharmacokinetics: measure of plasma colistimethate sodium, colistin A, and colistin B levels at multiple time points. Parameters: Cmax, AUC 0-t, Tmax, T1/2, Kel, clearance. Cohort 3 only. | Cohorts 3: Prior to first dose (less than and equal to 10 min); 30 minutes after the first dose in dosing periods 1 and 2; 30 minutes after the first IV and aerosol doses have both finished in dosing period 3
Pharmacokinetics: measure of plasma colistimethate sodium, colistin A, and colistin B levels at multiple time points. Parameters: Cmax, AUC 0-t, Tmax, T1/2, Kel, clearance. Cohort 4 only. | Cohorts 4: Prior to first dose (less than and equal to 10 min); 30 minutes after doses 7 and 13 in dosing period 1; 30 minutes after doses, 9 and 17 in dosing period 2; 30 minutes after doses 16 and 30 in dosing period 3
Pharmacokinetics: measure of plasma colistimethate sodium, colistin A, and colistin B levels at multiple time points. Parameters: Cmax, AUC 0-t, Tmax, T1/2, Kel, clearance. Cohorts 1-4. | Cohort 1-4: Prior to first dose (less than and equal to 10 min), immediately after (less than and equal to 10 min), 0.5, 1, 1.5, 2, 4, 8, 12 & 24 hours after the last dose in each dosing periods

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland
  - Case Western Reserve University - Case Medical Center - Infectious Disease & HIV Medicine, Cleveland, Ohio